CLINICAL TRIAL: NCT01294150
Title: Luminal Improvement Following Prostatic Tissue Approximation for the Treatment of Lower Urinary Tract Symptoms
Brief Title: The Safety and Effectiveness of UroLift: LIFT Pivotal Study
Acronym: LIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeoTract, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1012CP
Record Dates: First submitted 2011-02-07; First posted 2011-02-11 (Estimated); Results first posted 2015-08-13 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Cystoscopy; Cross-Over Studies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- UroLift System (Active Comparator): The treatment group subjects underwent the UroLift system procedure. The subject was blinded to his randomization into control or treatment group. Unblinding will occurred at 3 months post procedure after the assessments were completed. Between 3 and 12 month follow-up assessments, a subject was allowed to retreat with the UroLift system if he met the retreatment inclusion and exclusion criteria. Subjects that went on to UL retreatment within the first 12 months started their follow-up schedule over and were considered treatment failures. All UL subjects will be followed a minimum of 5 years.
  Interventions: Device: UroLift System
- Cystoscopy (Sham Comparator): The control group subjects underwent a cystoscopy procedure. The subject was blinded to his randomization into the control or treatment group. Unblinding will occurred at 3 months post procedure, after follow-up assessments were completed. Between 3 and 12 month follow-up assessments, a subject was allowed to crossover and undergo a UL procedure if he met crossover inclusion and exclusion criteria. Subjects crossing over will then be followed for 5 years post-treatment. The subject can also be treated by other approved therapies, or receive no treatment at all, which would require participation through 12 months.
  Interventions: Other: Cystoscopy
- Crossover (Active Comparator): Between 3 and 12 month follow-up assessments, a subject was allowed to crossover and undergo a UL procedure if he met crossover inclusion and exclusion criteria. Subjects crossing over will then be followed for 5 years post-treatment. The subject can also be treated by other approved therapies, or receive no treatment at all, which would require participation through 12 months.
  Interventions: Device: Crossover

INTERVENTIONS:
Device: UroLift System — The NeoTract UroLift System is a medical device approved for sale in the United States, European Union, and several other countries (see www.urolift.com). It was developed for the treatment of lower urinary tract symptoms (LUTS) associated with Benign Prostatic Hyperplasia (BPH). During the procedure, an implant is delivered into the prostatic lobe obstructing the urethra and restricting urine flow. The distal end of the device is used to compress the lobe then the implant is delivered to retain the lobe in position, thereby increasing the urethral opening and reducing the fluid obstruction through the prostatic urethra.
  Arms: UroLift System
Other: Cystoscopy — The Control Group will undergo cystoscopy.
  Arms: Cystoscopy
Device: Crossover — Subjects crossed over and received the UroLift System from the Control Group.
  Arms: Crossover

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of the UroLift(R) System when used in subjects with symptomatic benign hyperplasia (BPH). Primary effectiveness will be achieved by looking at the improvement of International Prostate Symptom Score (IPSS) and safety will be reviewed based on pertinent adverse events.

DETAILED DESCRIPTION:
The randomized portion of the study is a prospective, multicenter, multinational, 2:1 randomized, single-blinded controlled clinical trial comparing the IPSS of the treatment group to the IPSS of the control group at the 3 month follow-up. Subjects in the active treatment group undergo UroLift system treatment. Subjects in the control group undergo a cystoscopy procedure.

All subjects will be followed through 12 months, and through 5 years for those that receive the investigational device.

ELIGIBILITY:
Inclusion Criteria:

* Males age of 50 years or older diagnosed with symptomatic benign prostatic hyperplasia (BPH)

Exclusion Criteria:

* Size, volume,length of prostate

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2011-02; Primary Completion 2013-02 (Actual); Study Completion 2017-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claus Roehrborn, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (19):
- United States (14):
  - Genesis Research LLC, San Diego, California
  - Shahram S. Gholami MD - A Professional Corp., San Jose, California
  - Urology Associates of Denver, Englewood, Colorado
  - Advanced Urology Institute, Daytona Beach, Florida
  - Pinellas Urology, St. Petersburg, Florida
  - Northwestern University, Chicago, Illinois
  - Chesapeake Urology, Baltimore, Maryland
  - Sheldon J. Freedman, M.D., Ltd., Las Vegas, Nevada
  - Weill Cornell Medical College, New York, New York
  - Geisinger Medical Center, Danville, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - Scott and White Healthcare, Temple, Texas
  - Jean Brown Research, Salt Lake City, Utah
- Australia (3):
  - Figtree Private Hospital, Figtree, New South Wales
  - Austin Hospital, Heidelberg, Victoria
  - Port Macquarie Urology Centre, Port Macquarie
- Canada (2):
  - Oakville Trafalgar Memorial Hospital, Oakville, Ontario
  - Cam Am HIFU, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled into the L.I.F.T. clinical study on February 8, 2011. Study enrollment was completed on December 14, 2011 and the final subject reached the 12-month study endpoint on December 5, 2012.
Pre-assignment Details: Washout of for 3 months (5ARI) and 2 week (alpha blocker) required before baseline questionnaires.
Groups:
- UroLift System: The treatment group subjects underwent the UroLift (UL)system procedure. The subject was blinded as to whether he was in the control or treatment group. Unblinding occurred at 3 months post procedure after the assessments were completed. Between 3 and 12 month follow-up assessments, a subject was allowed to be retreated with the UroLift system if he met the retreatment inclusion and exclusion criteria. Subjects that went on to UL retreatment within the first 12 months were considered treatment failures, but started their follow-up schedule over. All subjects will be followed at a minimum of 5 years per the assessment schedule.
- Cystoscopy (Control/Sham): The control group subjects underwent a cystoscopy procedure. The subject was blinded as to whether he was randomized to the control or treatment group. Unblinding occurred at 3 months post procedure after follow-up assessments were completed. Between 3 and 12 month follow-up assessments, a subject was allowed to crossover and undergo procedure with the UroLift system, provided he met the inclusion and exclusion criteria. Subjects crossing over are then to be followed for 5 years post-treatment. If subject did not crossover, his participation was not required beyond the 12 month visit.
Period: Overall Study
Arm/Group | UroLift System | Cystoscopy (Control/Sham)
Started | 140 | 66
Completed | 138 | 64
Not Completed | 2 | 2
Not completed — Physician Decision | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- UroLift System: Average of 4.9 implants per prostate implanted. The prostatic urethral lift is performed by placing permanent transprostatic implants to lift apart the prostate lobes and reduce urethral obstruction.
- Cystoscopy: Sham treatment entailed rigid cystoscopy, a blinding screen and sounds that mimicked those of the prostatic urethral lift procedure.
- Total: Total of all reporting groups
Arm/Group | UroLift System | Cystoscopy | Total
Number analyzed (Participants) | 140 | 66 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (8.6) | 65 (8.0) | 66 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 140 | 66 | 206
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 136 | 63 | 199
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 3 | 5
  White | 131 | 62 | 193
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 94 | 45 | 139
  Canada | 20 | 10 | 30
  Australia | 26 | 11 | 37

OUTCOME MEASURES:

1. Primary Outcome: Collection of Post-treatment Catheterization for Safety
Description: The primary safety endpoint is an assessment of the rate of extended post-operative urinary catheterization in the subjects randomized to the UroLift group of the study in the ITT group. The extended post-operative urinary catheterization rate is defined as including those subjects who required catheterization within the first 3 days as part of post-operative management for inability to void, and required the catheter for more than 7 days. 2/140 met this endpoint.
Time Frame: Cath within first 3 days post-procedure which extended beyond 7 days, up to 12 days
Measure: Number; unit: participants
Groups:
- UroLift System: The treatment group subjects underwent UroLift system procedure. The subject was blinded to the randomization of control or treatment group. Unblinding occurred at 3 months post procedure after the assessments were completed. No matter which retreatment therapy, all subjects will be followed at a minimum of 5 years per the assessment schedule.
Arm/Group | UroLift System
Number analyzed (Participants) | 140
participants | 2

2. Primary Outcome: Comparison of IPSS for Efficacy
Description: The UroLift system will be considered superior to the Control if the mean International Prostate Symptom Score (IPSS) change (improvement) from baseline at 3 months demonstrates a minimum statistical margin of 25% compared to mean improvement from baseline for cystoscopy alone.
  The IPSS is an 8 question (7 symptom questions + 1 quality of life question) written screening tool used to screen for, rapidly diagnose, track the symptoms of, and suggest management of the symptoms of the disease benign prostatic hyperplasia (BPH).
  SCORING:
  0-7 Mildly symptomatic 8-19 Moderately symptomatic 20-35 Severely symptomatic
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: IPSS total score
Groups:
- UroLift System: The treatment group subjects underwent UroLift system procedure. The subject was blinded to the randomization of control or treatment group. Unblinding occurred at 3 months post procedure after the assessments were completed. All subjects will be followed at a minimum of 5 years per the assessment schedule.
- Cystoscopy: The control group subjects underwent a cystoscopy procedure only. The subject was blinded as to whether he was in the control or treatment group. Unblinding occurred at 3 months after follow-up assessments were completed. Between 3 and 12 month follow-up assessments, a subject was allowed to crossover and undergo the UroLift system procedure if he met inclusion and exclusion criteria. Subjects who crossed over will then be followed for 5 years post-treatment. The subjects that did not crossover were not required to participate beyond 12 months.
Arm/Group | UroLift System | Cystoscopy
Number analyzed (Participants) | 140 | 66
IPSS total score | 11.1 (7.67) | 5.9 (7.66)
Statistical Analysis 1: Comparison: UroLift System vs Cystoscopy; Test type: Superiority or Other; p = 0.003, t-test, 2 sided — Assuming unequal variances comparing mean improvement in the UL group to 125% of the mean improvement in the Control group. A p-value of 0.025 or less associated with UL is considered evidence of statistical significance

3. Primary Outcome: Mean UroLift Improvement in IPSS at 12 Months
Description: The International Prostate Symptom Score (IPSS) is a standardized 8 question (7 symptom questions + 1 quality of life question) written screening tool used to screen for, rapidly diagnose, track the symptoms of, and suggest management of the symptoms of the disease benign prostatic hyperplasia (BPH). Those patients scoring 7 or below are generally considered mildly symptomatic, whereas 20 or above is considered severely symptomatic. To meet co-primary effectiveness endpoint, the lower bound of a one-sided 97.5% confidence interval of IPSS mean percent change from baseline at Month 12 in the UroLift group must be greater than or equal to 30%.
Time Frame: 12 months
Measure: Number (97.5% Confidence Interval); unit: % IPSS Score Improvement
Arm/Group | UroLift System
Number analyzed (Participants) | 140
% IPSS Score Improvement | 45.5 [38.3 to NA] — This was a one-sided confidence interval

4. Secondary Outcome: Sexual Function
Description: Over the 12 month follow-up period, the proportion of UroLift patients who experience de novo sustained erectile dysfunction and retrograde ejaculation will be reported. Control subjects are not included in this analysis since controls could crossover option opened at 3 months.
Time Frame: 12 Months
Measure: Number; unit: % of Subjects
Arm/Group | UroLift System
Number analyzed (Participants) | 140
% of Subjects | 0.0

ADVERSE EVENTS:
Time Frame: Comparison safety data between two cohorts (we are listing 3 arms UroLift system, Cystoscopy and Crossover) at Index procedure through 5 Year Visit.
Description: All reported AEs are presented, including unrelated to device/procedure. The majority of the non-serious adverse events were deemed mild or moderate. No UADEs were reported through 5 Year Visit.
Groups:
- Crossover: Between 3 and 12 month follow-up assessments, a subject was allowed to crossover and undergo the UroLift system procedure if he met inclusion and exclusion criteria. Subjects who crossed over will then be followed for 5 years post-treatment. The subjects that did not crossover were not required to participate beyond 12 months.
Arm/Group | UroLift System | Crossover | Cystoscopy
All-Cause Mortality (participants affected / at risk) | 9/140 | 4/53 | 0/13
Serious Adverse Events (participants affected / at risk) | 52/140 | 19/53 | 0/13
Other Adverse Events (participants affected / at risk) | 133/140 | 49/53 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UroLift System (N=140) | Crossover (N=53) | Cystoscopy (N=13)
Haematuria (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) — Highly probable related to procedure and device
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) — cognard dural fistula
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Cardiac Arrythmia
Calculus urinary (Renal and urinary disorders) | 3 (3) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 1 (2) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Brain Hemorrhage
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery bypass (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) — Coronary artery disease
Coronary artery disease (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) — 1 = Shortness of breath
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) — Blood Clot in Right Leg
Dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — frontotemporal dementia
Embolism pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 1 (2) | 0 (0) | 0 (0) — Left Hip Replacement Right Hip Replacement
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — right hip fracture
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — ischemic cardiomyopathy related to class II heart failure
Joint arthroplasty (Surgical and medical procedures) | 1 (1) | 1 (2) | 0 (0) — right hip fracture
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — Recurrent renal cell carcinoma with metastasis
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — Metastatic Poorly Differentiated Squamous Cell Carcinoma
Myocardial infarction (Cardiac disorders) | 7 (7) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) — renal stone left side
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) — Diagnosis of pancreatic cancer
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Metastatic Pancreatic Cancer
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) — Peripheral vascular disease - Right lower limb
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Post-operative hemorrhage from a laparoscopic right inguinal hernia
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Renal cancer metastatic (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Residual urine (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Thyroid disorder (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Transient global amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Episode of apparent partial transient global amnesia
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transurethral prostatectomy (Surgical and medical procedures) | 3 (3) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Venous insufficiency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) — Chronic venous insufficiency - bilateral leg vein ligations
Whiplash injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — whiplash/headbump
Abscess (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Severe Right Carotid Artery Stenosis
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Fractured Nose
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) — Pinna Cancer
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — rt knee replacement
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) — mulitple myeloma with metastatic disease to bones
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Lumbar spondylosis
Testicular injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Epididymitis
Urine flow decreased (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Other, L2 Paraganglioma WHO grade 1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Coronary Arterial Stent Insertion (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UroLift System (N=140) | Crossover (N=53) | Cystoscopy (N=13)
Dysuria (Renal and urinary disorders) | 54 (57) | 21 (21) | 0 (0)
Haematuria (Renal and urinary disorders) | 47 (52) | 15 (15) | 0 (0)
Micturation Urgency (Renal and urinary disorders) | 20 (20) | 10 (11) | 0 (0)
Pelvic Pain (Renal and urinary disorders) | 28 (32) | 11 (12) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 21 (21) | 4 (4) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 10 (10) | 4 (4) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 19 (19) | 11 (11) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Nocturia (Renal and urinary disorders) | 10 (10) | 2 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 10 (10) | 5 (5) | 0 (0)
Prostatic specific antigen increased (Investigations) | 10 (10) | 5 (6) | 0 (0)
Residual urine (Renal and urinary disorders) | 7 (7) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 13 (15) | 8 (11) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator agreements restricted data disclosure until written agreement by or publication by Sponsor. The first publication appeared in the Journal of Urology, June 2013. "The Prostatic Urethral Lift for the Treatment of Lower Urinary Tract Symptoms Associated with Prostate Enlargement Due to Benign Prostatic Hyperplasia: The L.I.F.T. Study " Claus G. Roehrborn, Steven N. Gange, Neal D. Shore, Jonathan L. Giddens, et al. The Vol. 190, Issue 6, Pages 2161-2167.